CLINICAL TRIAL: NCT02088567
Title: A Prospective Randomized Clinical Trial Using Dehydrated Human Amnion/Chorion Membrane (dHACM) in Total Knee Replacement Patients to Reduce Post-operative Scarring.
Brief Title: Amniotic Membrane in Total Knee Replacements to Reduce Scarring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AFTKR001
Record Dates: First submitted 2013-11-21; First posted 2014-03-17 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Scarring
MeSH Terms: conditions — Cicatrix | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- dHACM (Experimental): Total knee arthroplasty, per the usual practice of the physician with application of dHACM between the underlying fascia and the overlying skin layers to reduce scar formation
  Interventions: Procedure: Total Knee Arthroplasty; Other: Application of dHACM
- Control (Other): Total knee arthroplasty, per the usual practice of the physician without application of dHACM.
  Interventions: Procedure: Total Knee Arthroplasty

INTERVENTIONS:
Procedure: Total Knee Arthroplasty — Total knee arthroplasty, per the usual practice of the physician.
Other: Application of dHACM — Application of dHACM at end of procedure before closing wound between the underlying fascia and the overlying skin layers to reduce scar formation
  Arms: dHACM

SUMMARY:
The overall objective of this study is to evaluate the effectiveness of dHACM in reducing scar tissue formation in total knee replacement patients.

ELIGIBILITY:
Inclusion Criteria:

1. Are adults ages 18 or older.
2. Are diagnosed with advanced osteoarthritis as determined by clinical exam and necessitate total knee replacement.
3. Have a willingness to comply with follow-up examination.
4. Have ability to give full written consent.

Exclusion Criteria:

1. Has had a previous total or partial joint replacement performed at the same site
2. Has a planned bilateral procedure at this time. Bilateral patients can be enrolled if the procedures are staged.
3. Has signs or symptoms of any other disease which could result in allograft failure, or has experienced allograft failure in the past.
4. Has used any investigational drug(s) or therapeutic device(s) within 30 days preceding screening.
5. Is pregnant or may become pregnant during the study.
6. Is a prisoner.
7. Has any condition(s) which seriously compromises the subject's ability to participate in this study, or has a known history of poor adherence with medical treatment.
8. Is currently taking medications which could affect allograft incorporation (supervising physician's discretion).
9. Is confined to bed or a wheelchair.
10. Has clinical signs and symptoms of local infection at the site.
11. Has autoimmune disease or a known history of having Acquired Immunodeficiency Syndrome (AIDS) or HIV.
12. Has current diagnosis of cancer at the site.
13. Has had prior radiation therapy treatment at the site.
14. Is currently taking anticoagulant therapy.
15. Is unable to sign or understand informed consent.
16. Has a history of drug or alcohol abuse within last 12 months.
17. Is allergic to Aminoglycoside antibiotics (such as gentamicin and/or streptomycin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Increased range of motion between both groups as measured by goniometer | 6 weeks

SECONDARY OUTCOMES:
Incidence of need for manual manipulation of affected knee | 6 weeks

OTHER OUTCOMES:
Increased Quality of Life as assessed by WOMAC and SF-36 | 6 weeks
  Western Ontario and McMaster Universities Arthritis Index (WOMAC) and Short Form 36 (SF-36) are measures of patient health status and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Jove, MD, Principal Investigator — Georgia Knee and Sports Medicine
Locations (1):
- Georgia Knee and Sports Medicine, Decatur, Georgia, United States